CLINICAL TRIAL: NCT05221541
Title: Is the Reflex Pathway Activated by Whole-body Vibration Change in Case of Voluntary Contraction?
Brief Title: Feature of Reflex Pathway Activated by WBV and Voluntary Contraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ilhan KARACAN, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TVRBMR
Record Dates: First submitted 2021-12-16; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Vibration; Exposure; Muscle Physiology
Keywords: muscle strength; vibration; reflex pathway
MeSH Terms: interventions — Vibration

STUDY DESIGN:
Intervention Model Description: Parallel group study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vibration (Experimental): Vibration (WBV and Tendon vibration) will be applied to participants
  Interventions: Procedure: vibration

INTERVENTIONS:
Procedure: vibration — whole-body vibration and soleus tendon vibration will be applied to participants

SUMMARY:
Whole-body vibration (WBV) has beneficial neuromuscular effects on muscle strength increase. Supraspinal, spinal, and peripheral mechanisms have been proposed to explain these beneficial effects. The most commonly proposed explanatory mechanism is spinal segmental reflexes. However, the neuronal circuit and receptors of the reflex response have not been defined precisely. A group of researchers found that the reflex system is the Tonic vibration reflex (TVR) under the neuromuscular effects of WBV; Other researchers claim that WBV activates a different spinal reflex than TVR.

Tonic vibration reflex is a polysynaptic reflex that occurs as a result of muscle spindle activation, in which more than 100 Hz vibrations are applied to the belly or tendon of the muscle.

A group of researchers argues that WBV activates the spinal reflex response, but this reflex response is different from TVR. According to them, WBV-induced reflex (WBV-IR) response latency is longer than TVR latency. WBV activates TVR at very attenuated amplitude; WBV activates a different spinal reflex with longer latency at medium and high amplitude vibration. They reported that although the H-reflex, T-reflex, and TVR latency was longer in the spastic soleus muscle than normotonic soleus muscle, where the muscle spindle and Ia afferent pathway were hyperactive. However, the WBV-IR latency was similar in both spastic and normotonic soleus muscle.

According to hypothesis of the present study , the reflex system activated by WBV changes depending on whether there is voluntary contraction or not: if the vibration is applied during voluntary contraction, the tonic vibration reflex is activated; In the absence of voluntary contraction (when the muscle is at rest), the bone myoregulation reflex is activated. The purpose of this research is to test this hypothesis.

DETAILED DESCRIPTION:
Subjects will be performed WBV in a semi-squatting position and standing upright, and soleus reflex latency will be detected by surface EMG during WBV. TVR latency will be measured by performing Achilles tendon vibration. Achilles tendon reflex latency will also be measured.

The WBV will be applied with the PowerPlate® Pro5 (London UK). The vibration amplitude will be 4 mm. The vibration frequency will be 30, 35, 40 Hz. Each vibration frequency will be applied for the 30s. A 10s rest period will be applied between vibrations of 30 seconds. This test vibration application will be performed in a semi-squatting position and standing upright. Subjects will be administered WBV for familiarisation prior to administration of WBV for testing purposes.

A surface EMG recording will be taken from the right soleus muscle belly. A pair of self-adhesive Ag/AgCl (KENDALL® Covidien, Massachusetts, USA) self-adhesive electrodes will have adhered to the skin. The surface EMG recordings will be made with a PowerLab ® (ADInstruments ADInstruments, Oxford, UK) data recorder with a sample rate of 40 kHz. EMG recordings will be analyzed offline with LabChart7 Pro® version 7.3.8 (ADInstruments, Oxford, UK).

For reflex latency calculation, piezo-electric accelerometers (LIS344ALH, ECOPACK®, Mansfield, TX, USA) will be fixed on the WBV device platform and on the right Achilles tendon. The acceleration data will be recorded with the PowerLab (ADInstruments London) data acquisition simultaneously with the EMG recording. Acceleration recording will be made with a sample rate of 40 kHz.

An electronic reflex hammer (Elcon, Germany) was used to determine T-reflex latency.

WBV-IMR and TVR latencies were then calculated by using the cumulative average method. All latencies were normalized to the body height of each participant. Latency was expressed as milliseconds (ms).

ELIGIBILITY:
Inclusion Criteria:

* Being healthy
* Being a young adult (20-45 years old)
* Volunteer

Exclusion Criteria:

* Scar, dermatitis, etc. in the skin tissue where the surface EMG electrode will be placed
* Kidney stone history
* Fracture in the lower extremity, history of orthopedic surgery
* Heart disease, Hypertension
* Dizziness
* Metabolic bone diseases, including osteoporosis
* History of bone occupying lesion, neoplasia, osteomyelitis
* Degenerative, inflammatory diseases of the joints of the lower extremities
* Lower extremity thrombophlebitis
* Lower extremity motor loss, sensory loss, muscle atrophy
* Subjects who cannot tolerate whole-body vibration

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
WBV-IR latency | 1 day
  Whole-body vibration induced reflex latency
TVR latency | 1 day
  Tonic vibration reflex latency
T-reflex latency | 1 day
  The Achilles tendon reflex latency

CONTACTS AND LOCATIONS:
Overall Officials: İLHAN KARACAN, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training & Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training & Research Hospital, Istanbul, Turkey (Türkiye)